CLINICAL TRIAL: NCT01797302
Title: Vitamin D and Vascular Function in Obese Children
Brief Title: Vitamin D and Vascular Health in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Kumaravel Rajakumar, Associate Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO12100034; R01HL112985 (NIH); 5R01HL112985-05 (NIH)
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Vitamin D Deficiency
Keywords: Obesity; Vitamin D Deficiency; Vascular Function; Insulin resistance; metabolic syndrome
MeSH Terms: conditions — Obesity; Vitamin D Deficiency; Insulin Resistance; Metabolic Syndrome | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vitamin D3 2000 IU (Active Comparator): Vitamin D3 2000 IU tablet once daily by mouth for 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3 1000 IU (Active Comparator): Vitamin D3 1000 IU tablet by mouth once daily for 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3 600 IU (Placebo Comparator): Vitamin D3 600 IU tablet by mouth once daily for 6 months
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Tablet form
  Other Names: Cholecalciferol

SUMMARY:
In this study, we will test the central hypothesis that enhancement of vitamin D status in obese and overweight children will improve their vascular health and their cardiovascular disease (CVD) and metabolic syndrome risk profile.

DETAILED DESCRIPTION:
Our primary objective is to determine, in obese and overweight children aged 10 to 18 years with vitamin D deficiency (defined as serum 25-hydroxyvitamin D <20 ng/mL), the efficacy of enhanced vitamin D3 supplementation in improving vascular endothelial function, arterial stiffness, insulin sensitivity, and metabolic syndrome risk status; and to assess whether these effects are dose-dependent. As a secondary objective, we will examine the vitamin D supplementation-induced effect on adipokines and inflammatory markers relevant to CVD risk. In a double-masked, controlled trial, we will randomize 252 eligible children to receive either 600 IU (conventional supplementation), or 1000 IU or 2000 IU (enhanced supplementation) of vitamin D3 daily for 6 months.

In terms of reporting of results, the following pre-specified outcomes are included in the primary manuscript (PubMed PMID:31950134 -- see Reference section for citation details)

1. Waist Circumference
2. Serum High Density Lipoprotein (HDL) Cholesterol
3. Serum Triglycerides
4. Inflammatory markers (Plasma TNF-alpha, high-sensitivity C-reactive protein, and IL-6)
5. Adiopkines (Plasma Leptin and Adiponectin)

Plasma nitric oxide metabolites were not measured.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be 10 to 18 years of age;
* obese or overweight (BMI ≥85th %tile);
* otherwise healthy, and
* have a serum 25(OH)D concentration <20 ng/mL

Children taking multivitamins should be able to hold off their multivitamins during the course of the study.

Exclusion Criteria:

Children will be excluded if they

* (a) have hepatic or renal disease, metabolic rickets, malabsorptive disorders, primary hyperparathyroidism, hyperthyroidism, or other chronic disorders that could affect vitamin D metabolism;
* (b) are receiving treatment with anticonvulsants, systemic glucocorticoids, pharmacologic doses of vitamin D (≥1000 IU of vitamin D2 or D3 daily), antihypertensives, vasoactive drugs, antilipidemics, metformin, antipsychotics, or other oral insulin regulators;
* (c) have cholelithiasis or urolithiasis;
* (d) have type 1 or type 2 diabetes; or
* (e) have a condition or underlying abnormality that could compromise the safety of the subject.

Post-menarchial girls with a positive pregnancy test at randomization, or subjects found during the screening phase to have hypercalcemia (serum calcium >10.8 mg/dL) or significant fasting hyperglycemia (fasting blood glucose ≥ 125 mg/dL) will also be excluded.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kumaravel Rajakumar, MD, MS, Principal Investigator — University of Pittsburgh, Children's Hospital of Pittsburgh of UPMC
Locations (1):
- Primary Care Center, Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Rajakumar K, Moore CG, Khalid AT, Vallejo AN, Virji MA, Holick MF, Greenspan SL, Arslanian S, Reis SE. Effect of vitamin D3 supplementation on vascular and metabolic health of vitamin D-deficient overweight and obese children: a randomized clinical trial. Am J Clin Nutr. 2020 Apr 1;111(4):757-768. doi: 10.1093/ajcn/nqz340. PMID 31950134

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Started | 75 | 74 | 76
3 Month Visit | 60 | 57 | 57
Completed | 58 | 48 | 50
Not Completed | 17 | 26 | 26
Not completed — Lost to Follow-up | 16 | 23 | 22
Not completed — Withdrawal by Subject | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU | Total
Number analyzed (Participants) | 75 | 74 | 76 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 (2.4) | 13.5 (2.2) | 13.5 (2.3) | 13.6 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 45 | 54 | 147
  Male | 27 | 29 | 22 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 2 | 10
  Not Hispanic or Latino | 68 | 73 | 74 | 215
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 70 | 70 | 71 | 211
  White | 11 | 12 | 8 | 31
  American Indian | 4 | 3 | 2 | 9
  Asian | 1 | 3 | 1 | 5
  Hawaiian | 0 | 0 | 1 | 1
  Other | 2 | 0 | 1 | 3
Body Mass Index [Mean (Standard Deviation); unit: "kg/m^2"] | 30.3 (5.8) | 30.0 (6.1) | 30.7 (6.9) | 30.3 (6.3)
Obese (BMI > or = 95th percentile) [Count of Participants; unit: Participants] | 47 | 50 | 53 | 150
Serum 25-hydroxyvitamin D (25[OH]D) [Mean (Standard Deviation); unit: ng/mL] | 14.2 (3.5) | 14.4 (3.4) | 14.3 (4.3) | 14.3 (3.7)
Serum parathyroid hormone (PTH) [Mean (Standard Deviation); unit: pg/mL] | 52.0 (19.9) | 45.7 (18.0) | 51.7 (20.6) | 49.8 (19.6)

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Dilation (FMD) Percentage
Description: Brachial artery flow-mediated dilation percentage is a measure of endothelial function. FMD percentage calculation is based on baseline brachial artery diameter(brachialADbase) and change in brachial artery diameter (brachialADchange) during post-occlusive reactive hyperemia. FMD% was determined using the formula (brachialADchange/brachialADbase) x 100.
Time Frame: 6 months
Population: Intention to treat with all available data
Measure: Mean (Standard Deviation); unit: percentage of baseline dilation
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 58 | 47 | 50
percentage of baseline dilation | 7.61 (5.15) | 8.27 (5.92) | 7.31 (5.14)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.88, Mixed Models Analysis — interaction term from model group*time

2. Secondary Outcome: Pulse-wave Velocity (PWV)
Description: PWV is a measure of arterial stiffness. Higher values of PWV indicate greater degree of arterial stiffness.
Time Frame: 6 months
Population: intention to tread with all available data
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 52 | 43 | 45
meters/second | 4.85 (0.76) | 4.85 (0.63) | 4.88 (0.75)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.85, Mixed Models Analysis — interaction term for group*time

3. Secondary Outcome: Augmentation Index at Heart Rate of 75 Beats/Min (AIx-75)
Description: AIx-75 is a measure of arterial stiffness. AIx was measured through radial arterial tonometry using SphygmoCor.
  Radial pulse waveform are analyzed through an automatic software function to determine aortic pulse waveform and aortic or central systolic (cSBP) and diastolic blood pressure (cDBP), and these measurements are further analyzed automatically to calculate AIx.
  AIx is a composite measure of the magnitude of wave reflection and arterial stiffness in all conduit arteries which affect the timing of the wave reflection. AIx = P2-P1/cSBP-cDBP, where P1 is the height of the incident pressure wave form during systole, P2 is the height of the reflected wave added to the incident wave, cSBP is the aortic systolic BP, and cDBP is the aortic diastolic BP. AIx adjusted to heart rate of 75 beats/min (AIx-75) is a validated index of arterial stiffness, with higher values indicating higher degree of arterial stiffness.
Time Frame: 6 months
Population: intention to treat with all available data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 57 | 46 | 44
ratio | 3.75 (8.44) | 2.22 (10.97) | 1.74 (10.29)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.61, Mixed Models Analysis — interaction term group*time from linear mixed model

4. Secondary Outcome: Central Systolic Blood Pressure
Description: a measure of cardiometabolic health
Time Frame: 6 months
Population: intention to treat with all available data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 57 | 46 | 44
mmHg | 98.45 (7.20) | 96.05 (8.19) | 98.50 (7.84)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.24, Mixed Models Analysis — interaction term group*time from linear mixed model

5. Secondary Outcome: Central Diastolic Blood Pressure
Description: a measure of cardiometabolic health
Time Frame: 6 months
Population: intention to treat with all available data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 57 | 46 | 44
mmHg | 68.69 (5.87) | 65.33 (8.27) | 68.57 (6.58)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.0117, Mixed Models Analysis — interaction term group*time from linear mixed model

6. Secondary Outcome: Systemic Systolic Blood Pressure
Description: a measure of cardiometabolic health
Time Frame: 6 months
Population: intention to treat with all available data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 58 | 48 | 50
mmHg | 114.71 (8.45) | 114.88 (11.76) | 115.70 (9.55)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.53, Mixed Models Analysis — interaction term group*time from linear mixed model

7. Secondary Outcome: Systemic Diastolic Blood Pressure
Description: a measure of cardiometabolic health
Time Frame: 6 months
Population: intention to treat with all available data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 58 | 48 | 50
mmHg | 67.57 (5.81) | 64.73 (8.44) | 67.30 (6.53)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.0256, Mixed Models Analysis — interaction term group*time from linear mixed model

8. Secondary Outcome: Fasting Blood Glucose
Description: a measure of cardiometabolic health
Time Frame: 6 months
Population: intention to treat with all available data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 58 | 48 | 50
mg/dL | 88.41 (6.33) | 88.48 (7.05) | 90.44 (6.04)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.0945, Mixed Models Analysis — interaction term group*time from linear mixed model

9. Secondary Outcome: 1/Fasting Insulin Ratio
Description: 1/fasting insulin ratio is a measure of insulin sensitivity. Increases in 1/fasting insulin ratio indicate improvements in insulin sensitivity.
Time Frame: 6 months
Population: intention to treat with all available data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 56 | 44 | 47
ratio | 0.08 (0.06) | 0.06 (0.04) | 0.06 (0.04)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.12, Mixed Models Analysis — interaction term group*time from linear mixed model

10. Other Pre Specified Outcome: Body Mass Index (BMI)
Description: a surrogate measure of adiposity
Time Frame: 6 months
Population: intention to treat with all available data
Measure: Mean (Standard Deviation); unit: "kg/m^2"
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
Number analyzed (Participants) | 58 | 48 | 50
"kg/m^2" | 30.82 (6.12) | 30.99 (6.41) | 30.62 (6.78)
Statistical Analysis 1: Comparison: Vitamin D3 2000 IU vs Vitamin D3 1000 IU vs Vitamin D3 600 IU; Test type: Superiority; p = 0.0094, Mixed Models Analysis — interaction term group*time from linear mixed model

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vitamin D3 2000 IU | Vitamin D3 1000 IU | Vitamin D3 600 IU
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/75 | 0/74 | 0/76
Other Adverse Events (participants affected / at risk) | 24/75 | 20/74 | 26/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 2000 IU (N=75) | Vitamin D3 1000 IU (N=74) | Vitamin D3 600 IU (N=76)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D3 2000 IU (N=75) | Vitamin D3 1000 IU (N=74) | Vitamin D3 600 IU (N=76)
Upper respiratory infection (Infections and infestations) | 9 (9) | 8 (8) | 8 (8)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Injury, poisoning, and proc complications other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous disorders other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures other (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Our findings of reductions in central-systolic BP and fasting glucose concentrations and improvement in insulin sensitivity lack adjustment for multiplicity and therefore should be considered as hypothesis-generating and interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT01797302/Prot_SAP_000.pdf